CLINICAL TRIAL: NCT00773331
Title: An Open Label Randomized Controlled Study to Compare the Efficacy and Safety of Once Every 4 Weeks Administration of Mircera Versus Short-acting Epoetin for the Maintenance of Hemoglobin Levels in Dialysis Patients With Chronic Renal Anemia.
Brief Title: A Study Comparing Maintenance of Hemoglobin Levels, Safety and Tolerability of Once Every 4 Weeks Mircera Versus Epoetin Beta in Dialysis Patients With Chronic Renal Anemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21904
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — epoetin beta; continuous erythropoietin receptor activator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]
- 2 (Active Comparator)
  Interventions: Drug: epoetin beta

INTERVENTIONS:
Drug: epoetin beta — As prescribed
  Arms: 2
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — 120, 200 or 360 micrograms every 4 weeks
  Arms: 1

SUMMARY:
This two arm study will compare the maintenance of hemoglobin levels, safety and tolerability of once every 4 weeks subcutaneous administration of Mircera versus epoetin beta in dialysis patients with chronic renal anemia. Patients will be randomized to receive either subcutaneous Mircera (starting dose 120, 200 or 360 micrograms) every 4 weeks or subcutaneous epoetin beta in accordance with the prescribed dosing information. In both groups, the starting dose will be the same as the previous dose of epoetin beta administered in the week preceding first study drug administration. Patients will be treated for 28 weeks with follow up 4 weeks after the last treatment visit. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* male or female patients, >=18 years of age;
* chronic renal anemia;
* Hb concentration 10.0 - 12.0 g/dL during the screening period;
* continuous subcutaneous maintenance therapy with epoetin at the same dose AND same dosing interval for at least 12 weeks before and throughout screening.

Exclusion Criteria:

* blood transfusion within the previous 8 weeks;
* poorly controlled hypertension;
* significant or acute or chronic bleeding;
* active malignant disease;
* congestive heart failure (NYHA Class IV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin concentration between baseline and the EEP | Week 20-28

SECONDARY OUTCOMES:
Proportion of patients maintaining average Hb concentration within the target range during the EEP; proportion of patients maintaining Hb concentration between 10-12g/dL throughout the EEP. | Weeks 1-28
Mean time spent in the Hb range 10 - 12g/dL; incidence of red blood cell transfusions during the DTP and EEP. | Weeks 1-28
Incidence of adverse events and serious adverse events; vital signs, laboratory parameters, ECG. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- China (6):
  - Beijing
  - Chengdu
  - Guangzhou
  - Hangzhou
  - Nanjing
  - Shanghai